CLINICAL TRIAL: NCT02158234
Title: A Phase I Dose Escalation Trial of Stereotactic Body Radiotherapy and Concurrent Cisplatin for Re-Irradiation of Unresectable, Recurrent Squamous Cell Carcinomas of the Head and Neck
Brief Title: Stereotactic Body Radiotherapy and Concurrent Cisplatin for Re-Irradiation of Unresectable, Recurrent Squamous Cell Carcinomas of Head and Neck
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-17799
Record Dates: First submitted 2014-06-04; First posted 2014-06-06 (Estimated); Last update posted 2023-01-19 (Actual); Status verified 2022-08

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: squamous cell carcinoma; head and neck cancer; paranasal sinuses; nasal cavity; nasopharynx; oropharynx; oral cavity; larynx; hypopharynx; salivary glands; cervical lymph nodes
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell; Head and Neck Neoplasms; Laryngeal Diseases | interventions — Cisplatin; Drug Therapy; Alkylating Agents; Radiosurgery; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation: SBRT and Cisplatin (Experimental): Stereotactic Body Radiation Therapy (SBRT) and Cisplatin. Starting Dose: 6 Gy/ Fraction 5/ Total 30 Gy/ Cisplatin 15 mg/m^2
  Interventions: Drug: Cisplatin; Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Drug: Cisplatin — Cisplatin 15 mg/m^2 prior to each fraction
  Other Names: chemotherapy; cis-diamminedichloroplatinum; CDDP; alkylating agent; cisplatinum
Radiation: Stereotactic Body Radiation Therapy (SBRT) — All participants will be treated every other day (excluding Saturday/Sunday). Starting Dose: 6 Gy/ Fraction 5/ Total 30 Gy.
  Other Names: stereotactic ablative radiotherapy; radiation therapy

SUMMARY:
This study involves another course of radiation (called re-irradiation) to the participant's tumor. The type of radiation is called stereotactic body radiation therapy (SBRT). The purpose of this study is to compare the effects, good and/or bad, of different doses of SBRT given along with the chemotherapy drug, cisplatin. The researchers want to see which dose of radiation will work best in controlling the growth of head/neck cancer. The usual treatment for head/neck cancer that has grown is surgery and/or more radiation with various chemotherapy drugs.

DETAILED DESCRIPTION:
Stereotactic Body Radiation Therapy (SBRT) is a relatively new radiation technique in which a few very high doses of radiation are delivered to small, well-defined tumors. It has been used effectively in other cancers like lung and liver. The goal is to deliver a radiation dose that is high enough to kill the cancer while limiting radiation to surrounding healthy organs. The daily dose of radiation is 2-3 times greater than conventional radiotherapy, but it is given for only 5 days over a 2 week period. Conventional radiotherapy is given over 6-7 weeks. The chemotherapy drug, cisplatin is used as a radiation sensitizer and will be given before each of the 5 radiation treatments.

ELIGIBILITY:
Inclusion Criteria:

* Recurrence of previously pathologically proven squamous cell carcinoma of the head and neck, including original primary sites in the paranasal sinuses, nasal cavity, nasopharynx, oropharynx, oral cavity, larynx, hypopharynx, salivary glands, and/or involvement of cervical lymph nodes
* Prior radiotherapy to doses ≥ 45 Gy to the area of recurrence, ≥ 6 months prior to enrollment
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 - 2
* Life expectancy > 6 months
* Medically unfit for surgery or deemed surgically unresectable by head and neck (H&N) surgeon within 60 days prior to enrollment, or patient refusal of surgery
* Normal organ and marrow function
* No prior evidence of Grade 3 or greater toxicity or neuropathy
* Medically fit to receive cisplatin

Exclusion Criteria:

* Positive urine pregnancy test and/or breastfeeding. Women of childbearing potential or sexually active males must be willing to use effective contraception throughout their participation in the treatment phase of the study.
* Evidence of distant metastases
* Tumor size > 7 cm in one direction
* Tumor within 1 cm of the spinal cord
* Cardiac history: class III or greater congestive heart failure (CHF) or myocardial infarction (MI) within last 6 months
* Medical condition or social situation that at the discretion of the principal investigator (PI) would preclude them from completion of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-07-16 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2021-08-24 (Actual)

PRIMARY OUTCOMES:
Maximal Tolerated Dose (MTD) of Stereoactive Body Radiation Therapy (SBRT) | Up to 24 months
  The traditional 3+3 dose escalation method will be utilized for this phase I study, with up to 3 sequential cohorts. The maximal tolerated dose (MTD) of Stereotactic Body Radiation Therapy (SBRT) radiation dose associated with a ≤ 33% probability of dose-limiting toxicity (DLT). DLT is defined as any grade 4 or greater toxicity, per The Common Terminology Criteria for Adverse Events v4 (CTCAE v4) that occurs within 3 months from the start of SBRT.

SECONDARY OUTCOMES:
Local Control Rate | Up to 24 months
  Local control is defined as lack of progression as defined radiographically or pathologically proven within the SBRT treated area. This will be calculated via Kaplan-Meier method. Response and progression will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) [Eur J Ca 45:228-247, 2009]. Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria.
Overall Survival (OS) | Up to 24 months
  Overall survival will be calculated from the end of SBRT treatment to time of death or last contact via Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Jimmy Caudell, M.D., Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States